CLINICAL TRIAL: NCT06082609
Title: Functional Relining Versus Digital Altered Cast Of Selective Pressure Impression Techniques Using Digitally Fabricated Distal Extension Frameworks: Abutment Alveolar Bone Height Changes
Brief Title: Functional Relining Versus Digital Altered Cast Using Digitally Fabricated Distal Extension Frameworks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Asmaa Sdeek, Principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A0104023RP
Record Dates: First submitted 2023-09-04; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Dental Prosthesis Complication
MeSH Terms: interventions — Denture, Partial, Removable

STUDY DESIGN:
Intervention Model Description: h. According to the functional impression techniques, all patients will be classified into two equal groups: Group A: Functional relining of processed RPD base at insertion Group B : Digitally obtained altered cast
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • Group 1 (Functional relining of processed RPD base at insertion) (Active Comparator): * After try in, a record base will be attached to the minor connectors and metal frameworks using 3D printed master cast.
  * Registration of jaw relation.
  * Mounting of master casts on articulator.
  * Setting of artificial teeth according to lingualized occlusion principles.
  * Try in of RPD.
  * Flasking of RPD to obtain mandibular distal extension removable partial dentures.
  * The finished removable partial denture is relined using the functional relining impression technique.
  Interventions: Procedure: Removable partial denture
- • Group 2 (Digitally obtained altered cast ); (Active Comparator): 1. Construction of custom tray on metal frame work.
  2. Border molding of custom tray.
  3. Selective pressure impression technique will be made.
  4. Digital altered cast will be done according to J. Wu, Y. Cheng
  5. 3D printing of altered master cast that will be used for completing the construction of RPD with the same steps of group (A) but without relining.
     * Finally the occlusion of dentures in the two groups will be verified before delivery.
  Interventions: Procedure: Removable partial denture

INTERVENTIONS:
Procedure: Removable partial denture — All patients will receive Removable partial denture by two different impression techniques

SUMMARY:
This clinical study will be done to compare between functional relining and digital altered cast of selective pressure impression techniques for constructing mandibular distal extension removable partial dentures using digitally fabricated frameworks by measuring the abutment alveolar bone height changes.

DETAILED DESCRIPTION:
According to the functional impression techniques, all patients will be classified into two equal groups:

Group A: Functional relining of processed RPD base at insertion:

•After try in, a record base will be attached to the minor connectors and metal frameworks using 3D printed master cast.The finished removable partial denture is relined using the functional relining impression technique.

Group B : Digitally obtained altered cast :

Selective pressure impression technique will be made.

Digital altered cast will be done according to J. Wu, Y. Cheng (20) as follow :

All patients will be informed about the follow up and evaluation recalls.

Evaluation of abutment alveolar bone height changes:

Alveolar bone height changes of abutment teeth will be evaluated radiographically at insertion (T0), and after 6 (T6) & 12 months (T12) after RPD insertion.

ELIGIBILITY:
Inclusion Criteria:

* 1. All patients having completely edentulous maxilla opposing class I Kennedy mandible.

  2. Sufficient restorative space must be available (from the mucosa covering the crest of the residual ridge to proposed occlusal plane). This will be detected by a tentative jaw relation.

  3. Well formed residual ridge covered by healthy firm mucosa. 4. All patients are of angel's class I maxillo-mandibular relationships. 5. Abutment teeth must fulfil certain criteria:
  1. Abutment teeth should be healthy with good periodontal and bone support.
  2. Should not show a pronounced degree of mobility or advanced gingival recession.
  3. Crown Root Ratio of abutment teeth not more than 1:2

     Exclusion Criteria:
* 1. Sever soft tissue undercuts. 2. Systemic diseases that may affect bone changes such as diabetes and osteoporosis.

  3. History of radiotherapy in the head and neck region.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
abutment alveolar bone loss | Two year
  Alveolar b(one height changes of abutment teeth will be evaluated radiographically at insertion and after one year

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University ,Faculty of dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No